CLINICAL TRIAL: NCT04184102
Title: The Impact of Therapeutic Exercises on the Quality of Life and Shoulder Range of Motion in Women After a Mastectomy, a Randomized Control Trial (RCT)
Brief Title: .Exercise and Follow-up After a Mastectomy
Acronym: mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NU04
Record Dates: First submitted 2019-10-23; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-10

CONDITIONS: Mastectomy; Lymphedema
Keywords: mastectomy; education; exercise
MeSH Terms: conditions — Lymphedema; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to a control of experimental group by flipping a coin
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention exercise (Experimental): The experimental group received education and exercise training before a mastectomy.
  Interventions: Behavioral: education
- Control (No Intervention): Received routine hospital care which did not include any exercise education

INTERVENTIONS:
Behavioral: education — The intervention group received pre-surgery education and training on therapeutic exercises in addition to the routine hospital care. The educational material was developed by the principal investigator (PI) and included a power point and a booklet with instructions on the exercises as well as information about the surgery and what to expect after the surgery. The educational material was based on previous research and adopted to our population after consultation with a panel of experts including two nurses and three physicians. Eligible women were approached while waiting for their appointment with their surgeon. If they showed interest in participating they signed a consent form. The PI explained the study and what is involved in participating including the weekly phone calls for women in the intervention group. Participants were told that they will visited at home by the PI to assess their ROM and to fill out a questionnaire.
  Other Names: Exercise Modeling
  Arms: Intervention exercise

SUMMARY:
A Randomized Control Trial (RCT) on the effect of education and Exercise on women after a mastectomy found positive results in range of motion of the affected shoulder and quality of life in the intervention group.

DETAILED DESCRIPTION:
Background: Breast cancer ranks highest in incidence and mortality among females and ranks second when both genders are combined. Lebanon has the second highest rate of breast cancer worldwide for the 35-39 age group and the highest in the 40-49 age group. Mastectomy often results in deceased shoulder and arm mobility, and decreased Quality of Life.

Objective: The objective of this study was to assess the effect of an educational program of therapeutic exercises on the quality of life and functional ability in women after a mastectomy Methods: Sixty women undergoing mastectomy were randomly assigned to an intervention and control group. The intervention group received extensive teaching pre-surgery education as well as training on therapeutic exercises. Follow up phone calls to the Intervention group were made to assure that the exercises were being done. Both groups were visited at home at four and eight to obtain the outcome variables. The Breast Cancer Patient Version was used to asses quality of life and the "Goniometer" was used to assess the range of motion of the affected shoulder.

ELIGIBILITY:
Inclusion criteria included:

* women between 35 and 55 years of age
* diagnosed with breast cancer
* scheduled for modified radical mastectomy. .

Exclusion Criteria included:

* Women who were pregnant,
* not able to communicate,
* had co-morbidities that affected their QoL

Ages: 33 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * women diagnosed with breast cancer
  * women undergoing a modified radical mastectomy
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Measuring the range of motion of the affected shoulder at two weeks. | At 2 weeks after surgery
  Measurement of shoulder range of motion using a Goniometer at two time points. The goniometer is a reliable tool which has been used in several studies to assess ROM of the of affected shoulder in patients after mastectomy. The goniometer assesses the range of motion, flexion, unbending, abduction, external rotation, and inward rotation of the shoulder joint. Normal values are abduction: 150 degrees. adduction: 30 degrees, orward flexion: 150-180 degrees, Extension: 45-60 degrees and rotation (test with elbow flexed to 90 degrees). The "Goniometer" is a nonintrusive and the most commonly used method to assess the ROM of a joint due to its simplicity and ease to implement The goniometer is a reliable tool which has been used in several studies to assess ROM of the of affected shoulder in patients after mastectomy.The goniometer assesses the range of motion, flexion, unbending, abduction, external rotation, and inward rotation of the shoulder joint.
Measuring the range of motion of the affected shoulder at four weeks. | At 4 weeks after surgery
  Measurement of shoulder range of motion using a Goniometer at two time points. The goniometer is a reliable tool which has been used in several studies to assess ROM of the of affected shoulder in patients after mastectomy. The goniometer assesses the range of motion, flexion, unbending, abduction, external rotation, and inward rotation of the shoulder joint. Normal values are abduction: 150 degrees. adduction: 30 degrees, orward flexion: 150-180 degrees, Extension: 45-60 degrees and rotation (test with elbow flexed to 90 degrees). The "Goniometer" is a nonintrusive and the most commonly used method to assess the ROM of a joint due to its simplicity and ease to implement The goniometer is a reliable tool which has been used in several studies to assess ROM of the of affected shoulder in patients after mastectomy.The goniometer assesses the range of motion, flexion, unbending, abduction, external rotation, and inward rotation of the shoulder joint.
Assessing the quality of life of participants at two weeks | At two weeks after surgery
  Qaulity of lfe was assessed at points in time. The Quality of Life Instrument: The Breast Cancer Patient Version (QoL-BC) was used to asses QoL. The QoL-BC is a patient self-reported scale assessing concerns of cancer survivors.It includes 46 items assessing four domains: 1) physical well-being (8 items), 2) psychological well-being, (22 items), 3) social well-being,(9 items) and 4) spiritual well-being (7 items). The itmes are scored form 0 to 10, 0 = worst outcome to 10 = best outcome. Several items have reverse anchors and therefore when you code the items you will need to reverse the scores of those items. Higher scores indicate better outocme.The overall and the subscales instrument have shown excellent internal and external reliability and moderate to strong validity.The QoL-BC has been translated to Arabic and used with breast cancer patients in several Arab countries with good reliability and validity.
Assessing the Quality of life of participants at four weeks | At 4 weeks after surgery
  Qaulity of lfe was assessed at points in time. The Quality of Life Instrument: The Breast Cancer Patient Version (QoL-BC) was used to asses QoL. The QoL-BC is a patient self-reported scale assessing concerns of cancer survivors.It includes 46 items assessing four domains: 1) physical well-being (8 items), 2) psychological well-being, (22 items), 3) social well-being,(9 items) and 4) spiritual well-being (7 items). The itmes are scored form 0 to 10, 0 = worst outcome to 10 = best outcome. Several items have reverse anchors and therefore when you code the items you will need to reverse the scores of those items. Higher scores indicate better outocme.The overall and the subscales instrument have shown excellent internal and external reliability and moderate to strong validity.The QoL-BC has been translated to Arabic and used with breast cancer patients in several Arab countries with good reliability and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Iman Kouatly, MpH, Study Director — American University of Beirut Medical Center
Locations (1):
- American University Medical Center (AUBMC), Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garlick M, Wall K, Corwin D, Koopman C. Psycho-spiritual integrative therapy for women with primary breast cancer. J Clin Psychol Med Settings. 2011 Mar;18(1):78-90. doi: 10.1007/s10880-011-9224-9. PMID 21344265
- [Background] Eyigor S, Karapolat H, Yesil H, Uslu R, Durmaz B. Effects of pilates exercises on functional capacity, flexibility, fatigue, depression and quality of life in female breast cancer patients: a randomized controlled study. Eur J Phys Rehabil Med. 2010 Dec;46(4):481-7. PMID 21224783
- [Background] Brandstatter M, Kogler M, Baumann U, Fensterer V, Kuchenhoff H, Borasio GD, Fegg MJ. Experience of meaning in life in bereaved informal caregivers of palliative care patients. Support Care Cancer. 2014 May;22(5):1391-9. doi: 10.1007/s00520-013-2099-6. Epub 2014 Jan 3. PMID 24382677
- [Background] Yildiz I, Varol U, Alacacioglu A. Assessment of the Quality of Life in Turkish Breast Cancer Patients. J Breast Health. 2014 Oct 1;10(4):216-221. doi: 10.5152/tjbh.2014.2012. eCollection 2014 Oct. PMID 28331674
- [Background] Sisman H, Sahin B, Duman BB, Tanriverdi G. Nurse-assisted education and exercise decrease the prevalence and morbidity of lymphedema following breast cancer surgery. J BUON. 2012 Jul-Sep;17(3):565-9. PMID 23033300
- [Background] Bluethmann SM, Vernon SW, Gabriel KP, Murphy CC, Bartholomew LK. Taking the next step: a systematic review and meta-analysis of physical activity and behavior change interventions in recent post-treatment breast cancer survivors. Breast Cancer Res Treat. 2015 Jan;149(2):331-42. doi: 10.1007/s10549-014-3255-5. Epub 2015 Jan 3. PMID 25555831
- [Background] McNeely ML, Campbell K, Ospina M, Rowe BH, Dabbs K, Klassen TP, Mackey J, Courneya K. Exercise interventions for upper-limb dysfunction due to breast cancer treatment. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD005211. doi: 10.1002/14651858.CD005211.pub2. PMID 20556760
- [Result] Benton MJ, Schlairet MC, Graham HL. Physical activity-related quality of life in breast cancer survivors compared to healthy women. Eur J Cancer Care (Engl). 2019 Nov;28(6):e13142. doi: 10.1111/ecc.13142. Epub 2019 Aug 29. PMID 31465139
- [Derived] Majed M, Neimi CA, Youssef SM, Takey KA, Badr LK. The Impact of Therapeutic Exercises on the Quality of Life and Shoulder Range of Motion in Women After a Mastectomy, an RCT. J Cancer Educ. 2022 Jun;37(3):843-851. doi: 10.1007/s13187-020-01894-z. Epub 2020 Nov 20. PMID 33219500

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT04184102/Prot_SAP_000.pdf